CLINICAL TRIAL: NCT01851070
Title: A Double-blind, Randomized, Placebo-controlled, Dose-escalation, Multi-center Study a Single Intravenous Infusion of Allogeneic Mesenchymal Precursor Cells (MPCs) in Patients With Rheumatoid Arthritis and Incomplete Response to at Least One TNFα Inhibitor
Brief Title: A Multi-center Study a Single IV Infusion of Allogeneic MPCs in Patients With Rheumatoid Arthritis and Incomplete Response to at Least One TNFα Inhibitor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mesoblast, Ltd. (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MSB-RA001
Record Dates: First submitted 2013-04-19; First posted 2013-05-10 (Estimated); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal Saline Placebo (Placebo Comparator): Placebo will be delivered in 100 mL normal saline administered intravenously over approximately 45 minutes.
  Interventions: Drug: Allogeneic Mesenchymal Precursor Cells
- Allogeneic Mesenchymal Precursor Cells (Active Comparator): Mesenchymal Precursor Cells (MPCs), either 1.0 or 2.0 million cells/kg, will be delivered in 100 mL normal saline administered intravenously over approximately 45 minutes.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Allogeneic Mesenchymal Precursor Cells
  Arms: Normal Saline Placebo
Drug: Normal Saline
  Arms: Allogeneic Mesenchymal Precursor Cells

SUMMARY:
Study is a double-blind, randomized, placebo controlled, dose escalating study. The primary objective of this study is to evaluate the safety, tolerability and feasibility of a single intravenous infusion of allogeneic mesenchymal precursor cells (MPCs) compared to placebo at 12 weeks post-infusion in the treatment of patients with active rheumatoid arthritis (RA) who have received methotrexate +/- other DMARDs for at least 6 months prior to screening and who have had an incomplete response to at least one TNF-alpha inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females ages 18-80 years old
* Active rheumatoid arthritis (RA) disease as per 2010 ACR/EULAR classification criteria for the diagnosis of RA.
* Must be positive for rheumatoid factor and/or anti-cyclic citrullinated peptide (anti-CCP3) but without extra-articular disease or functional limitation
* Patient with active RA defined as:

  * ≥ 4 tender joint count (TJC) 28 joint count at screening and
  * ≥ 4 swollen joint count (SJC) count 28 joint count at screening
  * ESR ≥ 28 mm/hr or hsCRP >2.0 mg/L
* Patient has been taking MTX for at least 4 months with dose and route of administration stable for at least 8 weeks prior to screening
* Patient has had an inadequate response to at least one TNFα inhibitor with last dose at least 6 weeks prior to screening
* Use of oral DMARD (sulfasalazine, hydroxychloroquine, chloroquine and leflunomide) is permitted but must be stable for at least 3 months prior to screening

Exclusion Criteria:

* Pregnant women or women who are breastfeeding.
* Other investigational therapy received within 8 weeks or five half-lives (whichever is longer) prior to Screening (except as in exclusion #13).
* Known or suspected alcohol or drug abuse within three years preceding Screening.
* Autoimmune disease other than RA (such as systemic lupus erythematosus (SLE), mixed connective tissue disease, scleroderma, polymyositis/dermatomyositis, vasculitis)
* History of or current inflammatory joint disease other than RA (such as tophaceous gout, reactive arthritis, psoriatic arthritis, ankylosing spondylitis or other spondyloarthropathy, Lyme disease). Patients primarily diagnosed with osteoarthritis are excluded.
* Bedridden or confined to a wheelchair or patients with > 3 arthroplasties due to RA.
* History of diagnosed and/or treated malignancy with no evidence of recurrence in past 5 years
* Surgical procedures planned to occur during the trial (these patients may be rescreened following completion of and recovery from the surgical procedure).
* Use of TNFα inhibitor for treatment of RA at time of screening or within the 6 weeks prior to screening.
* Prior use of biologic agent for treatment of RA within 6 weeks prior to screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of the safety of a single IV infusion of allogeneic MPCs compared to placebo at 12 weeks post-infusion | 12 weeks post IV Infusion
  To evaluate the safety, tolerability and feasibility of a single intravenous (IV) infusion of allogeneic mesenchymal precursor cells (MPCs) compared to placebo at 12 weeks post-infusion in the treatment of patients with active rheumatoid arthritis (RA) who have received methotrexate +/- other oral DMARDs for at least 4 months and who have had an incomplete response to at least one course of a TNFα inhibitor.
  Overall safety will be based on the overall assessment of AE/SAEs, Vital Signs, Physical Examination, clinical laboratory tests, ECGs and Chest x-ray.

SECONDARY OUTCOMES:
Evaluation of the efficacy of a single intravenous infusion of allogeneic MPCs compared with placebo at 12 weeks post-infusion with MPCs or placebo in the treatment of patients with active RA | 12 weeks post IV infusion with MPCs
  To assess the efficacy of a single intravenous infusion of allogeneic MPCs compared with placebo at 12 weeks post-infusion with MPCs or placebo in the treatment of patients with active RA who have received methotrexate +/- other DMARDs for at least 4 months and who have had an incomplete response to least one TNFα inhibitor.
Evaluation of long-term safety and efficacy of a singly IV infusion of allogeneic MPCs in patients with active RA | 52 weeks post IV Infusion
  To evaluate the long-term efficacy and safety of allogeneic MPCs over the entire study duration in the treatment of patients with active RA who have received methotrexate +/- other DMARDs for at least 4 months and who have had an incomplete response to at least one TNFα inhibitor
  Safety will be assessed according to the following:
  * Adverse events/serious adverse events ("primary endpoint")
  * Vital signs
  * Physical examination
  * Clinical laboratory tests
  * Electrocardiogram
  * Chest x-ray (CXR)
  Efficacy will be assessed according to the following:
  * ACR20/50/70
  * DAS28 (mean changes from baseline as measured by using hsCRP and ESR)
  * Mean changes from baseline in all components of the ACR core response criteria
  * Remissions (as defined in the 2011 Joint Statement of the American College of Rheumatology (ACR) and European League Against Rheumatism (EULAR)
  * Joint erosion of hands and wrists assessed via x-ray
  * Patient-reported outcomes
    * SF36v2
    * HAQ_DI

CONTACTS AND LOCATIONS:
Overall Officials: Donna Skerrett, MD, MS, Study Director — Mesoblast, Ltd.
Locations (23):
- United States (20):
  - Pinnacle Research Group, Anniston, Alabama
  - Arthrocare Arthritis Care and Research PC, Gilbert, Arizona
  - Triwest Research Associates, El Cajon, California
  - UCLA, Los Angeles, California
  - Inland Rheumatology Clinical Trials Incorporated, Upland, California
  - Ocala Rheumatology Research Center, Ocala, Florida
  - Arthritis Center, Palm Harbor, Florida
  - Sarasota Arthritis Research Center, Sarasota, Florida
  - McIlwain Medical Group, Tampa, Florida
  - JHU Arthritis Center Baltimore, Baltimore, Maryland
  - Arthritis Treatment Center, Frederick, Maryland
  - Reliant Medical Group, Worcester, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Office of Ramesh C. Gupta, MD, Fair Lawn, New Jersey
  - DJL Clinical Research, Charlotte, North Carolina
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - West Tennessee Research Institute, Jackson, Tennessee
  - Accurate Clinical Research, Houston, Texas
  - Texas Arthritis Research Center, San Antonio, Texas
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Southern Clinical Research Pty Ltd, Hobart, Tasmania
  - Emeritus Research, Malvern, Victoria